CLINICAL TRIAL: NCT06783257
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group Phase II Clinical Trial to Evaluate the Efficacy and Safety of Vonoprazan Fumarate Injection for the Treatment of Peptic Ulcer Bleeding
Brief Title: Phase II Clinical Study of Vonorasan Fumarate Injection in the Treatment of Peptic Ulcer Bleeding
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTP-FNLS-004
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Peptic Ulcer Bleeding
MeSH Terms: conditions — Peptic Ulcer Hemorrhage | interventions — Esomeprazole; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vonora fumarate Injections 1 (Experimental): 40 mg (20 mg bid, 6 hours apart, Day1) + 20 mg (Day2&3, q24h), ivd, 30 min, administered for 3 days
  Interventions: Drug: Vonorasan fumarate injection1
- Vonora fumarate Injections 2 (Experimental): 40mg（Day1）+20mg（Day 2&3），ivd，30min，q24h，administered for 3 days
  Interventions: Drug: Vonorasan fumarate injection2
- Esomeprazole sodium for injection (Active Comparator): 80mg，iv，30±3min； Followed by 8 mg/h, ivd, 71.5 h
  Interventions: Drug: Esomeprazole sodium for injection

INTERVENTIONS:
Drug: Vonorasan fumarate injection1 — 40 mg (20 mg bid, 6 hours apart, Day1) + 20 mg (Day2&3, q24h), ivd, 30 min, administered for 3 days
  Arms: Vonora fumarate Injections 1
Drug: Vonorasan fumarate injection2 — 40mg（Day1）+20mg（Day 2&3），ivd，30min，q24h，administered for 3 days
  Arms: Vonora fumarate Injections 2
Drug: Esomeprazole sodium for injection — 80mg，iv，30±3min； Followed by 8 mg/h, ivd, 71.5 h
  Arms: Esomeprazole sodium for injection

SUMMARY:
A Multicenter, Randomized, Double-Blind, Parallel-Group Phase II Clinical Trial to Evaluate the Efficacy and Safety of Vonoprazan Fumarate Injection for the Treatment of Peptic Ulcer Bleeding

DETAILED DESCRIPTION:
The trial was divided into screening period, treatment period and follow-up period.Subjects who did not meet the exclusion criteria were randomly assigned to vonorasan fumarate injection or esoprazole sodium for injection for 3 days; Safety was followed up to 2 days after the end of intravenous administration.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign the informed consent form.
2. Individuals aged between 18 and 75 years, regardless of gender.
3. Clinical manifestations of upper gastrointestinal bleeding, such as hematemesis, melena, or positive fecal occult blood, within 48 hours prior to screening.
4. Patients diagnosed with upper gastrointestinal bleeding caused by gastric and/or duodenal ulcers through endoscopic examination within 24 hours prior to random group selection, with ulcer maximum diameter ranging from 3 to 20 mm.
5. The classification of peptic ulcers according to Forrest is as follows: Ia, Ib, IIa, IIb. For multiple ulcers, the higher Forrest grade is used for determination. After confirming the ability to achieve hemostasis through endoscopic treatment, the following requirements for endoscopic treatment are as follows:

   * For Forrest Ia, Ib, IIa: Thermal hemostasis or mechanical hemostasis is the primary method, and it is also permissible to combine local epinephrine injection based on the aforementioned primary methods;
   * For Forrest IIb: To confirm the specific grade, endoscopic irrigation to remove attached blood clots should be attempted first. If the blood clots are cleared, the Forrest grade should be reassessed. If it is classified as Forrest Ia, Ib, or IIa, endoscopic hemostatic treatment should be performed as per the above requirements. If the blood clots are not cleared and it is ultimately confirmed as Forrest IIb, direct grouping is permitted.

Exclusion Criteria:

1. Individuals with a clinically significant history of drug allergies or known allergies to the components and excipients of the study drug;
2. Subjects with other severe central nervous system, cardiovascular, respiratory, organ, renal, gastrointestinal, urinary, endocrine, or hematological diseases, which the investigator believes may confound the study results or affect the safety of the subjects;
3. Hematological disorders: ① Platelet count <80×10^9/L; ② PT exceeds the upper limit of normal by 3 seconds; ③ APTT exceeds the upper limit of normal by 10 seconds; (If any of these criteria are met, the patient is not eligible for selection)
4. Renal function abnormalities: ① ALT or AST ≥1.5×ULN; ② Total bilirubin >1.5×ULN; ③ Serum creatinine (Cr) > ULN; (If any of these criteria are met, the patient is not eligible for selection)
5. A history of drug abuse within the last 5 years;
6. Receipt of live vaccines or attenuated live vaccines within 30 days prior to the first administration, or plans to receive vaccinations during the study period;
7. Hemorrhagic shock (occurring during the screening period with systolic blood pressure <90 mmHg and heart rate >120 beats/min, accompanied by symptoms such as pallor, cold and clammy extremities, restlessness, or altered mental status) or requiring arterial catheter embolization or surgical intervention due to unsuccessful endoscopic treatment;
8. Concurrent upper gastrointestinal bleeding from other causes or suspected gastric malignancy under endoscopy; There is a clear history of surgery to reduce gastric acid or a history of gastric surgery (including but not limited to partial gastrectomy, gastric plasty, vagotomy, excluding simple perforation suturing);

10. A history of malignant tumors within 5 years prior to screening (if the subject has been cured of skin basal cell carcinoma or cervical carcinoma in situ, he/she may participate in this study); 11. Use of proton pump inhibitors (PPIs) or H2 receptor antagonists or P-CAB preparations exceeding a single dose of the standard dose within 24 hours prior to screening, or having undergone endoscopic treatment/intervention before signing the informed consent form, and having used PPIs, P-CAB preparations, H2 receptor antagonists, somatostatin, or hemostatic agents after endoscopic treatment/intervention until the selection for this study; 12. Patients currently using drugs with a clear risk of interaction with the investigational drug, such as azanavir sulfate, nelfinavir, saquinavir, or liponavir; 13. Use of hemostatic powder Endoclot AHP® or other local hemostatic agents during endoscopy that, in the investigator's judgment, affect the efficacy of the investigational drug; 14. Pregnant or breastfeeding women, as well as those with plans for pregnancy or sperm/egg donation within 3 months after the end of the study, who are unwilling to adopt a medically recognized contraceptive method (such as an intrauterine device or condom) during the study; 15. Participation in other drug/device clinical studies and use of investigational drugs/devices within 3 months prior to randomization; 16. Other subjects deemed unsuitable for selection by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The rebleeding rate within 72 hours after the initiation of medication evaluated by endoscopy. | 72 hours

SECONDARY OUTCOMES:
The rebleeding rate within 72 hours and 120 hours after the initiation of medication clinical evaluation. | 72 hours, 120 hours
The transfusion rate and average transfusion volume of subjects due to bleeding within 72 hours and 120 hours after the initiation of medication; | 72 hours, 120 hours
The proportion of subjects who required re-endoscopic hemostatic treatment due to bleeding within 72 hours and 120 hours after the initiation of medication. | 72 hours, 120 hours
The proportion of subjects who required surgical treatment due to bleeding within 72 hours and 120 hours after the initiation of medication. | 72 hours, 120 hours
The mortality rate of subjects within 72 hours and 120 hours after the initiation of medication. | 72 hours, 120 hours
The incidence ofadverse reactions | 120 hours